CLINICAL TRIAL: NCT03616860
Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier Disruption for the Treatment of High Grade Glioma in Patients Undergoing Standard Chemotherapy
Brief Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier (BBB) Disruption for Treatment of Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT008C; 277981 (Other: Health Canada)
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Focused Ultrasound (FUS) BBB Disruption (Experimental): The Exablate Model 4000 Type 2 system is intended for use as a tool to induce localized and temporary blood-brain barrier disruption in patients with glioblastoma undergoing standard of care chemotherapy.
  Interventions: Device: Focused Ultrasound (FUS) BBB Disruption

INTERVENTIONS:
Device: Focused Ultrasound (FUS) BBB Disruption — FUS BBB disruption involves the application of acoustic energy at low frequencies from over 1000 individual transducers into distinct body targets
  Other Names: Exablate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety of blood-brain barrier (BBB) disruption in adult patients with a first presentation of a glioblastoma (GBM) following a maximal safe surgical resection and standard chemo-radiation with temozolomide (TMZ) protocol and ready for the maintenance phase of the Stupp protocol with TMZ.

DETAILED DESCRIPTION:
This is a prospective, single center, single-arm study to establish the safety, feasibility, and effectiveness of BBB disruption along the periphery of the tumor resection cavity using the ExAblate Neuro Model 4000 Type 2 (220 kHz) system and DEFINITY ultrasound contrast in patients with GBM. Adult patients with a first time diagnosis of GBM, whom have undergone maximal safe surgical resection and have safely completed the initial phase of concurrent chemo-radiation therapy, will be recruited for this study. Twenty patients will undergo up to 6 treatments with FUS coincident with their standard TMZ cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women.
2. Age between 18 and 80 years, inclusive.
3. Able and willing to give informed consent.
4. Grade IV malignant glioma (GBM) confirmed through assessment of surgical specimens by a board-certified neuropathologist.
5. Undergone maximal safe surgical resection and completed concurrent radiotherapy+oral TMZ without any complications and deemed eligible for the maintenance phase of TMZ treatment.
6. Karnofsky rating 70-100.
7. ASA score 1-3.
8. Able to communicate during the ExAblate MRgFUS procedure.
9. Able to attend all study visits (i.e., life expectancy of at least 3 months).

Exclusion Criteria:

1. Patients presenting with the following imaging characteristics:

   i. Evidence of recent intracranial hemorrhage.
2. The sonication pathway to the tumour involves:

   i. Extensive scalp scars, ii. Clips or other metallic implanted objects in the skull or the brain (brain implants).
3. The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema).
4. Patients requiring increasing doses of corticosteroids.
5. Patient receiving bevacizumab (Avastin) therapy.
6. Patients undergoing other concurrent therapies such as chemotherapy wafers, immunotoxins delivered by convection-enhanced delivery, regionally administered gene and viral therapies, immunotherapies, and focal irradiation with brachytherapy, stereotactic radiosurgery, and laser interstitial thermotherapy.
7. Cardiac disease or unstable hemodynamics including:

   i. Documented myocardial infarction within six months of enrollment. ii. Unstable angina on medication. iii. Congestive heart failure. iv. Left ventricular ejection fraction <50%. v. History of a hemodynamically unstable cardiac arrhythmia. vi. Cardiac pacemaker.
8. Severe hypertension (diastolic BP > 100 on medication).
9. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment.
10. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumour hemorrhage.
11. Documented cerebral infarction within the past 12 months.
12. TIA in the last 1 month.
13. Cerebral or systemic vasculopathy.
14. Insulin-dependent diabetes mellitus that is not well-controlled or that in the Investigator's opinion precludes participation in the study.
15. Known sensitivity to gadolinium-DTPA.
16. Known sensitivity to DEFINITY ultrasound contrast agent or perflutren.
17. Contraindications to MRI such as non-MRI-compatible implanted devices.
18. Large subjects not fitting comfortably into the MRI scanner.
19. Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia.
20. Untreated, uncontrolled sleep apnea.
21. Positive pregnancy test (for pre-menopausal women).
22. Known life-threatening systemic disease.
23. Severely impaired renal function.
24. Cardiac shunt.
25. Previous full course of chemotherapy.
26. Allergy to eggs or egg products.
27. Subjects with evidence of cranial or systemic infection.
28. Subjects with chronic pulmonary disorders.
29. Subjects with a history of drug allergies, asthma or hay fever, and multiple allergies, in particular subjects with a history of anaphylaxis.
30. Subjects with evidence of Hepatitis B virus infection/carrier state.
31. Liver injury as indicated by liver function tests.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Device and procedure related adverse events | Throughout the study, approximately 12 months.
  The number and severity of device and BBB disruption procedure related adverse events will be evaluated and classified according to the CTCAE

SECONDARY OUTCOMES:
Feasibility of repeated BBB disruption will be evaluated through assessment of post-procedure contrast-enhanced magnetic resonance (MR) imaging | Immediately after each FUS BBB disruption procedure
  The repeatability of BBB disruption will be evaluated at each of the 6 procedures (coincident with standard of care chemotherapy) and will be evaluated through assessment of post-procedure contrast enhanced MR imaging.
Effectiveness of BBB disruption in the treated tumor region | at each standard of care neuro-oncology follow up visit until date of death from any cause, assessed up to 48 months
  Effectiveness will be assessed based on the MRI characteristics of the FUS treated tumor region as assessed by the modified Response Assessment in Neuro-Oncology Criteria (RANO) to establish GBM status

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodworth GF, Anastasiadis P, Ozair A, Chabros J, Bettegowda C, Chen C, Gerstl JVE, Douville C, Mekary RA, Smith TR, Meng Y, Hawkins C, Pople CB, Abrahao A, Llinas M, Heyn C, Bunevicius A, Rezai AR, Ball AJS, Henry K, Sahgal A, Torio E, Ren H, Ahmad H, Arora H, Eisenberg H, Perry J, Carpenter JS, Hynynen K, Pham LC, Anketell MB, Lim-Fat MJ, Xu Z, Cifarelli CP, Sheehan JP, McDannold NJ, Gandhi D, Golby AJ, Lipsman N. Microbubble-enhanced transcranial focused ultrasound with temozolomide for patients with high-grade glioma (BT008NA): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2025 Dec;26(12):1651-1664. doi: 10.1016/S1470-2045(25)00492-9. PMID 41308679
- [Derived] Meng Y, Pople CB, Suppiah S, Llinas M, Huang Y, Sahgal A, Perry J, Keith J, Davidson B, Hamani C, Amemiya Y, Seth A, Leong H, Heyn CC, Aubert I, Hynynen K, Lipsman N. MR-guided focused ultrasound liquid biopsy enriches circulating biomarkers in patients with brain tumors. Neuro Oncol. 2021 Oct 1;23(10):1789-1797. doi: 10.1093/neuonc/noab057. PMID 33693781